CLINICAL TRIAL: NCT01352208
Title: Phase I/II, Multi-center, Open Label, Study to Assess the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Anti Tumor Activity of ASP9521 in Patients With Metastatic Castrate-resistant Prostate Cancer
Brief Title: Phase I/II Study of ASP9521 in Castrate-Resistant Prostate Cancer (CRPC) Patients
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: It was decided to discontinue the development in consideration of the results of a P1 study
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9521-CL-0002; 2010-023382-22 (EudraCT Number)
Record Dates: First submitted 2011-04-14; First posted 2011-05-11 (Estimated); Last update posted 2014-03-24 (Estimated); Status verified 2012-12

CONDITIONS: Castrate Resistant Prostate Cancer
Keywords: ASP9521; Castrate Resistant Prostate Cancer; Phase 1/2
MeSH Terms: interventions — 1-(1-((5-methoxy-1H-indol-2-yl)carbonyl)piperidin-4-yl)-2-methylpropan-2-ol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ASP9521 (Experimental)
  Interventions: Drug: ASP9521

INTERVENTIONS:
Drug: ASP9521 — oral

SUMMARY:
The study has three parts. Part 1 is a dose escalation to investigate the safety and tolerability of ASP9521. Part 2 will evaluate the safety and tolerability and initial anti-tumor activity of ASP9521. Part 3 of the study will be a Food Effect study.

DETAILED DESCRIPTION:
The purpose of the first study part is to investigate the safety and tolerability of ASP9521 in patients with Castrate Resistant Prostate Cancer. This will be done at different doses, starting at the lowest dose up to higher doses to find the maximum dose that is tolerated.

The second part will investigate the safety and tolerability and evaluate initial anti-tumor activity of ASP9521. This will be done at multiple doses which are identified in part 1 to potentially be effective. The number of patients in part 2 will be higher number compared to part I.

The third part of the study will investigate the effect of food on the drug in patients; this will be a crossover design fed to fasted and vice versa.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate without neuroendocrine differentiation or small cell features
* Metastatic disease documented by 2 or more bone lesions on bone scan or by soft tissue disease observed by Computed tomography/Magnetic resonance imaging (CT/MRI)
* Ongoing androgen deprivation with Luteinizing hormone-releasing hormone (LHRH) agonist/antagonist therapy or bilateral orchiectomy. For patients who have not had an orchiectomy, there must be a plan to maintain effective LHRH agonist/antagonist therapy for the duration of the study
* Serum testosterone <1.7 nmol/L (50 ng/dL) at screening
* Patients receiving bisphosphonates or other approved bone targeting therapy must have been on stable doses for at least 4 weeks prior to screening
* Progressive disease at study entry defined as one or more of the following 3 criteria occurring in the setting of castrate levels of testosterone:

  * Prostate-specific antigen (PSA) progression defined by a minimum of 2 rising PSA levels with an interval of >1 week between each determination. The PSA value at screening should be >2 ng/mL
  * Soft tissue disease progression defined by Response Evaluation Criteria in Solid Tumors (RECIST). Measurable disease is not required for entry. Lymph nodes >20 mm are considered measurable disease
  * Bone disease progression defined by at least 2 new lesions on bone scan
* Life expectancy of >6 months according to the investigator's judgment
* Chemotherapy-Naïve patients should be asymptomatic or controlled symptomatic patients with metastatic CRPC who have failed one or more lines of hormonal treatment/androgen deprivation therapy but have not received chemotherapy or have refused chemotherapy. Post chemotherapy patients should have received not more than two prior regimens of chemotherapy for prostate cancer, of which one is docetaxel-based

Exclusion Criteria:

* Concomitant treatment with the following is prohibited:

  * All biologic agents (except for sipuleucel T [Provenge®]), or other agents with anti-tumor activity against prostate cancer, including 5 alpha reductase inhibitors, androgens (e.g., testosterone), cytoproterone acetate and all other progestational agents, estrogens, and flutamide within 4 weeks prior to screening
  * Bicalutamide or nilutamide within 6 weeks prior to screening
  * Treatment with estramustine
  * Ketoconazole for treatment of prostate cancer
  * Treatment with abiraterone
* Radiation therapy for treatment of the prostate within 3 months prior to screening
* Radiation therapy for the treatment of metastases within 3 weeks (if single fraction of radiotherapy then within 2 weeks) and radionuclide therapy for the treatment of metastases within 4 weeks prior to screening
* Major surgery within 2 months prior to screening
* Known or suspected intracerebral disease or brain metastasis
* Use of an investigational agent within 4 weeks prior to treatment allocation or a period required by local regulation, whichever is longer
* Prior use, or participation in a clinical study, of an investigational agent that blocks androgen synthesis or targets the androgen receptor

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2011-03; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability, based on the frequency and severity of Adverse Events (AEs), laboratory assessments, vital signs, electrocardiograms (ECGs) and clinical observations | Up to day 28 and further

SECONDARY OUTCOMES:
Decline in Prostate-specific antigen (PSA) | Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Director — Astellas Pharma Europe B.V.
Locations (4):
- Site 131, Antwerp, Belgium
- Site: 121, Villejuif, France
- United Kingdom (2):
  - Site:109, Glasgow
  - Site: 101, Surrey

REFERENCES:
- [Derived] Loriot Y, Fizazi K, Jones RJ, Van den Brande J, Molife RL, Omlin A, James ND, Baskin-Bey E, Heeringa M, Baron B, Holtkamp GM, Ouatas T, De Bono JS. Safety, tolerability and anti-tumour activity of the androgen biosynthesis inhibitor ASP9521 in patients with metastatic castration-resistant prostate cancer: multi-centre phase I/II study. Invest New Drugs. 2014 Oct;32(5):995-1004. doi: 10.1007/s10637-014-0101-x. Epub 2014 Apr 27. PMID 24771350